CLINICAL TRIAL: NCT00273949
Title: Lactulose for the Prevention of Nosocomial Infections in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: BZ00001
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2008-02-06 (Estimated); Status verified 2005-09

CONDITIONS: Nosocomial Infection
Keywords: Lactulose; Prebiotics; Nosocomial infection; children; infants
MeSH Terms: conditions — Cross Infection | interventions — Lactulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: lactulose

SUMMARY:
The purpose of this study is to assess the ability of lactulose, a prebiotic agent, to prevent hospital acquired infection in children

DETAILED DESCRIPTION:
Despite the adoption of norms regarding enteric isolation, nosocomial infectious diarrhea is common in children(1;2). Viral pathogens, especially rotavirus are responsible for most of the cases. Depending on population, type of hospital, and standard of care, the reported incidence rate ranges from 8 to 33 episodes per 100 admissions(1). Infants and toddlers are at the highest risk of acquiring nosocomial viral gastroenteritis(1;2).

Probiotic bacteria have been shown to be beneficial in the prevention and treatment of gastrointestinal infections as well as reduction of viral shedding(3;4). A recent study by Szajewska et al. (2) showed a significant reduction of nosocomial infections from 33% to 7% by prophylactic treatment with LGG during the hospital stay. Another study however, did not show any difference(1).

Another approach is to use prebiotic treatment. Prebiotics are defined as non-digestible substances that, when ingested, selectively promote the growth and establishment of beneficial probiotic-like bacteria normally present in the gut(5).

Lactulose is a semi-synthetic disaccharide made from lactose by a chemical reaction which was first described in 1930(6).

In contrast to other prebiotics, lactulose has up to now been mainly used as a medicinal drug for constipation and hepatic encephalopathy(6). In 1957 Petuely published the basic work about lactulose as "the bifidus factor" which was confirmed by MacGillivray et al(6).They found that the composition of the colonic microflora of bottle-fed babies is very much like that of adults while if lactulose is added to the formula milk such babies have the same composition as breast-fed babies.

Lactulose has been used for 40 years in the treatment of constipation [10] and for more than 30 years for encephalopathy.The dosages used in PSE are up to four times higher than those usually applied in constipation. No putative or definite evidence of mutagenic, genotoxic or teratogenic effects of lactulose has been obtained in human use. Animal studies in rats and rabbits also did not reveal any teratogenic or reproduction-toxicologic effects, and even high dosages have had no deleterious effects(6)

Our hypothesis is that lactulose, with its proven prebiotic properties, given to children during their hospital stay, would be beneficial in reducing nosocomial infections.

ELIGIBILITY:
Inclusion Criteria:

* All children aged 2 to 36 months who are admitted to the hospital for reasons other than diarrhea will be eligible for the study.

Exclusion Criteria:

* Children with a history of probiotics or prebiotics use within 7 days before admission, acute gastroenteritis within 3 days before admission, vomiting, treated chronic constipation, known anatomic problem in the gastrointestinal tract will be excluded from the study.

Ages: 2 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100
Dates: Start 2006-01; Study Completion 2007-01

PRIMARY OUTCOMES:
The incidence of diarrhea

SECONDARY OUTCOMES:
Incidence of rotavirus diarrhea

CONTACTS AND LOCATIONS:
Overall Officials: Ron Shaoul, Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Pediatric Department, Bnai Zion Medical Center, Haifa, Israel

REFERENCES:
- [Background] Mastretta E, Longo P, Laccisaglia A, Balbo L, Russo R, Mazzaccara A, Gianino P. Effect of Lactobacillus GG and breast-feeding in the prevention of rotavirus nosocomial infection. J Pediatr Gastroenterol Nutr. 2002 Oct;35(4):527-31. doi: 10.1097/00005176-200210000-00013. PMID 12394379
- [Background] Szajewska H, Kotowska M, Mrukowicz JZ, Armanska M, Mikolajczyk W. Efficacy of Lactobacillus GG in prevention of nosocomial diarrhea in infants. J Pediatr. 2001 Mar;138(3):361-5. doi: 10.1067/mpd.2001.111321. PMID 11241043
- [Background] Schumann C. Medical, nutritional and technological properties of lactulose. An update. Eur J Nutr. 2002 Nov;41 Suppl 1:I17-25. doi: 10.1007/s00394-002-1103-6. PMID 12420112